CLINICAL TRIAL: NCT06694857
Title: 3-Dimensional Volumetric Analysis of a Hyaluronic Filler Injection for Jaw Contouring
Brief Title: A Prospective Evaluation of the Filler for Jaw Contouring
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Principal Investigator, Ivona Percec, Associate Director, Cosmetic Surgery, University of Pennsylvania
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB#855232
Record Dates: First submitted 2024-11-15; First posted 2024-11-19 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Dermal Fillers
Keywords: Jaw; Hyaluronic Acid; HA Filler; Hyaluronic Acid Filler; Filler; Cosmetic; Face; Dermal Fillers; Chin
MeSH Terms: conditions — Facies

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Filler (Experimental): HA Filler to jaw line
  Interventions: Drug: HA filler

INTERVENTIONS:
Drug: HA filler — patient will receive FDA approved dosages of filler to the lower face region to treat facial contour or asymmetry, as per FDA approved indications. Patients are limited to 20 mL of any JUVÉDERM® injectable gel per 60 kg (132 lbs) body mass per year. Prior to injection patients will be imaged with 3-dimensional photogrammetry. Subjects will return post-injection in 2 weeks, 1 month, and 3 months for re-imaging.

SUMMARY:
The goal of this prospective study is to analyze volumetric changes in the lower face after hyaluronic acid filler injections over 90 days. The main question it aims to answer is:

To quantify volume change of the lower face area over time after injection of filler

* Participants will receive hyaluronic acid filler injections (Juvéderm Volux XC) for contouring of the jawline. Each patient will receive FDA approved dosages of filler to the lower face region to treat facial contour or asymmetry, as per FDA approved indications.
* Prior to injection patients will be imaged with 3-dimensional photogrammetry. Subjects will return post-injection in 2 weeks, 1 month, and 3 months for re-imaging.

ELIGIBILITY:
Inclusion Criteria:

1. Age 22-55
2. Patients interested in jaw contouring
3. Participants must sign the informed consent form.

Exclusion Criteria:

1Prior filler for facial contouring 2) Filler injection within the past 12 months or during duration of study 3) Prior facial cosmetic surgery (ie. facelift) 4) Prior facial trauma (ie. orbital fracture) 5) Pregnant or breastfeeding 6) Planned dental work within next 2 weeks 7) The following contraindications: patients with severe allergies manifested by a history of anaphylaxis or history or presence of multiple severe allergies, gram-positive bacterial protein allergies and lidocaine allergies

Ages: 22 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2024-10-31 (Actual); Primary Completion 2025-11-01 (Actual); Study Completion 2025-11-01 (Actual)

PRIMARY OUTCOMES:
Volume change of the lower face area at 30 days post-intervention | 30 days
  3D- images will be collected to determine change in volume following from pre-intervention to post-intervention (30 days)

SECONDARY OUTCOMES:
PRO | 90 Days
  Determine patient satisfaction with lower face volume changes as determined by PROs via Validated FACE-Q Aesthetics questionnaire. Scale scores range from 0 (lowest) to 100 (highest).
Volume Change of the Lower Face 14 days Post-intervention | 14 days
  3D- images will be collected to determine change in volume following from pre-intervention to post-intervention (14 days)
Volume changes of the lower face at 90 days post-intervention | 90 days
  3D- images will be collected to determine change in volume following from pre-intervention to post-intervention (90 days)

CONTACTS AND LOCATIONS:
Locations (1):
- Penn Medicine, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No